CLINICAL TRIAL: NCT03060798
Title: The Change of Tissue Oxygen Saturation Measured by Dynamic Near Infrared Spectroscopy Following Volatile Anesthesia in Healthy Population
Brief Title: The Change of Tissue Oxygen Saturation Following Volatile Anesthesia
Status: Completed | Type: Observational
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Hyeon-Jeong Lee, Associate Professor, Pusan National University Hospital
Other Study IDs: 1607-012-054
Record Dates: First submitted 2017-02-19; First posted 2017-02-23 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Healthy; Aging
MeSH Terms: interventions — Desflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Drug: Desflurane — general anesthesia using desflurane.
  Other Names: suprane
Device: Near-infrared spectroscopy monitor — tissue oxygen saturation monitoring combined with vessel occlusion test
  Other Names: tissue oxygen saturation monitor

SUMMARY:
General anesthesia can affect tissue oxygen saturation and microcirculatory reactivity. However, the differences in microcirculation caused by anesthetic methods have not been well studied. Near-infrared spectroscopy (NIRS) measures peripheral tissue oxygen saturation noninvasively and can be used in conjunction with vascular occlusion (VOT) experiments. The purpose of this study was to examine the changes in NIRS derived tissue oxygen saturation (StO2) and microcirculatory reactivity by VOT after inhalation anesthesia in healthy population.

This prospective, observational study will be performed on 60 healthy patients who had undergone elective surgery under volatile general anesthesia. The investigators measure StO2 and microvascular reactivity using NIRS combined with vascular occlusion test (VOT). The parameters were performed twice per patient, before and after the induction of anesthesia.

Occlusion slope and recovery slope during VOT will be compared before and after anesthesia. Moreover, the changes depend on the age will be analyzed.

DETAILED DESCRIPTION:
This prospective observational study was performed on 60 patients without comorbidities who underwent elective surgery under general anesthesia. Before and after the induction of anesthesia, StO2 monitoring and VOT were performed to investigate the effect of anesthesia on microcirculation. To investigate the effect of age on microcirculation, the patients were divided into two different groups, young (< 65 yrs) and old (> 65 yrs) groups, and the VOT-derived parameters and hemodynamics between two groups were compared.

ELIGIBILITY:
Inclusion Criteria:

* Adult Over 18 years of age undergoing general surgery under general anesthesia.

Exclusion Criteria:

* ASA category III or IV, Diabetes, Chronic Kidney Disease, Vascular Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male and female patients over 18 years of age undergoing general surgery under general anesthesia. American anesthesiologists association patient (ASA) category I or II.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in Tissue Oxygen Saturation after General Anesthesia | before and 30 minutes after anesthetic induction
  Vascular occlusion test (VOT) will be performed twice for each patient, before (T0) and 30 min after the induction of general anesthesia (T1). Before induction, a NIRS sensor will be placed on the thenar eminence and an automated tourniquet will be placed around the ipsilateral upper arm. After the baseline StO2 stabilization, the automatic tourniquet will be inflated to 50 mmHg over the patient's baseline systolic blood pressure and maintain for 5 min. After the 5-min ischemic period, the tourniquet will be rapidly deflated to 0 mmHg. StO2 data will be continuously recorded during the VOT procedure. Baseline StO2, minimum StO2 during the 5-min inflation of the tourniquet, maximum StO2 during deflation of the tourniquet, time to minimum StO2, and time to maximum StO2 will be obtained. The occlusion slope and recovery slope will be calculated based on the measured StO2 data.

SECONDARY OUTCOMES:
Age-related changes in microcirculation | before and 30 minutes after anesthetic induction
  Patients will be divided into three groups by age (younger group: < 65 years old and older group: ≥ 65 years old) to perform age-based analysis. The acquired StO2 data by the VOT test among the groups will be analyzed and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon-Jeong Lee, PhD, Principal Investigator — Pusan National University Hospital
Locations (1):
- Hyeon Jeong Lee, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No